CLINICAL TRIAL: NCT00001320
Title: I-123 Iodobenzamide (IBZM) SPECT Studies of D2 Receptor Distribution and Function in Patients With Schizophrenia and Normal Volunteers
Brief Title: Neuroimaging of Dopamine Metabolism in Normal and Psychiatric Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920024; 92-M-0024
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-07

CONDITIONS: Healthy; Schizophrenia
Keywords: Parkinson's Disease; Schizophrenia; Dopamine D2/D3 receptors; Brain Imaging; SPECT; Equilibrium; Brain Scan; Brain Research; Brain Disorders; Schizoaffective Disorder; Normal Volunteer
MeSH Terms: conditions — Schizophrenia; Parkinson Disease; Brain Diseases; Psychotic Disorders

SUMMARY:
Brain cells communicate with each other by releasing chemicals called neurotransmitters. In order for brain cells to transfer information, one cell will release a neurotransmitter that will be recognized by a receptor located on surface of another cell. One such neurotransmitter is dopamine.

Abnormal dopamine transmission has been seen in patients with substance abuse and different neuropsychiatric disorders including schizophrenia.

A radioactive drug called IZBM (I-123 iodobenzamide) can also bind to certain dopamine receptors. IZBM can be seen by Single Photon Emission Tomography (SPECT). Therefore, by using IZBM and SPECT scans, researchers can find and "map" the location of dopamine receptors in the brain.

Patients participating in this study must also have been selected for other genetic studies being conducted at the NIMH. Patients with schizophrenia will be selected from a NIMH research study titled, "Neurobiological Investigation of Patients with Schizophrenia Spectrum Disorders and Their Siblings" (95-M-0150). Normal patient volunteers will be selected from another NIMH study titled, "Inpatient Evaluation of Neuropsychiatric Patients" (89-M-0160). All aspects of clinical care and genetic analysis of these patients will be covered in these studies, while information pertaining to IBZM SPECT scans will be covered in this study.

This study will not directly benefit patients participating in it. However, information gathered may contribute to faster and more accurate diagnosis of schizophrenia and eventually better treatment for the disorder.

DETAILED DESCRIPTION:
Abnormalities in dopaminergic neurotransmission have been described in substance abuse and different neuropsychiatric disorders including schizophrenia. [I-123] IBZM is a radioligand that has been widely employed for SPECT imaging of dopamine type 2 and type 3 receptors (D2 and D3, respectively) and fluctuations in levels of endogenous dopamine. [I-123] IBZM SPECT has been used in the SPECT Lab of the Clinical Brain Disorders Branch for several years without adverse effects. Pharmacological effects of IBZM are unlikely due to the minimal amounts used and have not been observed. We propose to use [I-123] IBZM SPECT to explore following questions: 1) Can a previously found relationship between N-acetylaspartate (NAA) measures in the dorsolateral prefrontal cortex and striatal dopamine activity in patients with schizophrenia be replicated and is it also found in normal subjects? 2) Do allelic variants of genes for the dopamine type 2 (DRD2) and type 3 (DRD3) receptors, the dopamine transporter (SLC6A3), or enzymes involved in dopamine biosynthesis (TH) and metabolism (COMT, MAOA) affect D2 receptor availability in vivo?

This technical protocol describes the procedural aspects of [I-123]IBZM SPECT. It is not intended to be sufficient on its own for a clinical study. All subjects volunteering for this study will be recruited from among individuals who have previously consented to participate in clinical studies under one of two NIH protocols that include genetic testing. Schizophrenia patients will be recruited from among NIMH inpatients participating under NIH protocol #89-M-0160, "Inpatient Evaluation of Neuropsychiatric Patients" (Egan 1999a). Normal volunteers will be recruited from among those participating under NIH protocol #95-M-0150, "A Neurobiological Investigation of Patients with Schizophrenia Spectrum Disorders and Their Siblings" (Egan 1999b), which includes recruitment of a normal control group whose first degree relatives are free of mental illness. All details related to clinical care and genetic analysis are contained in those two protocols and their associated consent forms; all details related to [I-123]IBZM SPECT studies, per se, are discussed in this protocol, which requires a separate informed consent from each volunteer.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with schizophrenia will be recruited exclusively from among inpatients who are participating in clinical studies of the Clinical Brain Disorders Branch of NIMH under NIH protocol #89-M-0160 (Egan 1999a) and for whom genetic data is already available.

Normal volunteers will be recruited exclusively from among individuals who have volunteered for studies under NIH protocol #95-M-0150 (Egan 1999b) as normal control subjects and for whom genetic data is already being analyzed.

EXCLUSION CRITERIA:

Pregnancy: All women of childbearing age must undergo a pregnancy test prior to injection or radioactive isotope. If the pregnancy test is positive or if the woman has reason to believe she might be pregnant, she will be excluded from this study.

Breastfeeding: Women who are breastfeeding will be excluded from this study to avoid unwarranted risk to their children.

Iodine sensitivity: Subjects with a prior reaction to iodine, iodine compounds, or shellfish will be excluded from this study. Also, subjects with a history of thyroid disease or dysfunction will be excluded from this study.

Substance abuse: Subjects with a history of recent substance abuse will be excluded from this study.

Metal objects in body: Subjects with metal objects in their bodies as specified in our MRI protocol (91-M-0124) will be excluded from this study.

INCLUSION CRITERIA FOR PATIENTS WITH SCHIZOPHRENIA:

Prior participation as a NIMH inpatient under NIH protocol #89-M-0160.

Schizophrenia diagnosis according to DSM-IV criteria.

EXCLUSION CRITERIA FOR PATIENTS WITH SCHIZOPHRENIA:

Coexistence of another mental illness at the time of the study. If the patient has experienced other mental illnesses in the past (e.g. a learning disability or major depression), then this should be judged to be fully recovered.

INCLUSION CRITERIA FOR NORMAL CONTROLS:

Prior participation as a normal volunteer under NIH protocol #95-M-0150.

No Axis I or Axis II diagnoses.

EXCLUSION CRITERIA FOR NORMAL CONTROLS:

Subjects with an Axis I or II disorder will be excluded.

Subjects with concomitant medical or neurological disorders which require ongoing medication, or which may affect the central nervous system will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 265
Dates: Start 1991-10; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Knable MB, Egan MF, Heinz A, Gorey J, Lee KS, Coppola R, Weinberger DR. Altered dopaminergic function and negative symptoms in drug-free patients with schizophrenia. [123I]-iodobenzamide SPECT study. Br J Psychiatry. 1997 Dec;171:574-7. doi: 10.1192/bjp.171.6.574. PMID 9519100
- [Background] Knable MB, Heinz A, Raedler T, Weinberger DR. Extrapyramidal side effects with risperidone and haloperidol at comparable D2 receptor occupancy levels. Psychiatry Res. 1997 Sep 29;75(2):91-101. doi: 10.1016/s0925-4927(97)00023-1. PMID 9351491
- [Background] Wolf SS, Jones DW, Knable MB, Gorey JG, Lee KS, Hyde TM, Coppola R, Weinberger DR. Tourette syndrome: prediction of phenotypic variation in monozygotic twins by caudate nucleus D2 receptor binding. Science. 1996 Aug 30;273(5279):1225-7. doi: 10.1126/science.273.5279.1225. PMID 8703056